CLINICAL TRIAL: NCT03973073
Title: Evaluation of the Potential Interference of Camouflage on the Treatment of Vitiligo: an Observer-blinded Self-controlled Study
Brief Title: Effects of Combination Therapy With Camouflage in the Repigmentation of Vitiligo
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, dujuan, chief physician of dermatology, Principal investigator, clinical professor, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2019PHB002-01
Record Dates: First submitted 2019-06-02; First posted 2019-06-04 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Vitiligo
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- camouflage group (Experimental): Topical applications and/or NB-UVB plus Capulin TM on-demand treatment period
  Interventions: Combination Product: CapulinTM; Other: topical applications and NB-UVB
- blank group (Other): Topical applications and/or NB-UVB on-demand treatment
  Interventions: Other: topical applications and NB-UVB

INTERVENTIONS:
Combination Product: CapulinTM — camouflage
  Arms: camouflage group
Other: topical applications and NB-UVB — combination therapy of vitiligo

SUMMARY:
Vitiligo is a common depigmented skin disorder characterized by the white patches of skin and mucous membrane. It can be cosmetically disfiguring and lead to serious psychological problems for patients with vitiligo. In view of the difficulty of vitiligo treatment, the combination therapy is the most recommended. Despite that, the process of repigmentation usually last for several months to several years. So it is of great value to explore therapeutic methods that can improve appearance, relieve patients' pain and improve their quality of life in the process of treatment. The use of camouflage can vastly improve quality of life, both the European and Japanese guidelines of vitiligo management recommend that once vitiligo is diagnosed, camouflage should be used. The first commercial camouflage agent in China is CapulinTM by 2004. The main component of it is dihydroxyacetone. The repigmented mechanism is to combine with the keratin and to form a special brown polymer, which makes leukoderma close to normal skin. While, it is unknown whether camouflage has an impact on the drug absorption, efficiency of phototherapy and thus influences the repigmentation of vitiligo. Thus, the investigators undergo a randomized open-label self-controlled study to estimate the effects of combination therapy between camouflage and topical application and/or NB-UVB in the repigmentation of vitiligo.

DETAILED DESCRIPTION:
Vitiligo is a common depigmented skin disorder characterized by the white patches of skin and mucous membrane. It can be cosmetically disfiguring and lead to serious psychological problems for patients with vitiligo, especially when the exposed skin are involved, such as face and extremities.

The pathogenesis of vitiligo is not clear yet. The most common methods of treatment include systemic corticosteroids, topical application (such as corticosteroids, calcineurin inhibitors), phototherapy, traditional medications and so on. In view of the difficulty of vitiligo treatment, the combination therapy between drugs and phototherapy is the most recommended. Despite that, the process of repigmentation usually last for several months to several years. So it is of great value to explore therapeutic methods that can improve appearance, relieve patients' pain and improve their quality of life in the process of treatment.

For patients seeking to mask their vitiligo, camouflage options have historically been limited and been designated as a cosmetic, rather than a medical concern. As research has indicated that proper concealment of vitiligo lesions can vastly improve quality of life, we believe it is essential that dermatologists become aware of all the options available to their patients and that discussions of camouflage options be broached from the first visit. Until now, both the European and Japanese guidelines of vitiligo management recommend that once vitiligo is diagnosed, camouflage should be used.

The first commercial camouflage agent in China is CapulinTM by 2004. The main component of CapulinTM is dihydroxyacetone, and it also contains natural plant extracts, moisturizers, emollients and natural pigments. The repigmented mechanism is to combine with the keratin and to form a special brown polymer, which makes leukoderma close to normal skin.

Although the guidelines of home and abroad consider camouflage as the fundamental treatment of vitiligo, it is unknown whether camouflage has an impact on the drug absorption, efficiency of phototherapy and thus influences the repigmentation of vitiligo.

Thus, the investigators undergo a randomized observer-blinded self-controlled study to estimate the effects of combination therapy between camouflage and topical application and/or NB-UVB in the repigmentation of vitiligo.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who signed Informed Consent Form；
* Male or female subjects 16 years of age or older；
* Clinically confirmed diagnosis of vitiligo；
* Existing 2 symmetrical or adjacent white patches with similar size or a single lesion area greater than 5 cm2

Exclusion Criteria:

* Tend to automatically repigment；
* Allergic history of any relevant ingredient in the camouflage;
* The combination of eczema, contact dermatitis, urticaria and other allergic diseases or other serious diseases which are not suitable for the treatment of skin diseases；
* Women of child-bearing potential who are pregnant, plan to become pregnant during study or are lactating；
* Any other condition that the investigator deems unsuitable for entering the study.

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-21 (Actual)

PRIMARY OUTCOMES:
Repigmentation area of vitiligo | 12 weeks
  The primary endpoint was percentage of repigmentation, assessed using photographs taken at baseline and each follow up visit. The photographs were shown to three dermatologists (blinded observers) for independent assessment and a mean of these values was taken.

SECONDARY OUTCOMES:
types of regimentation types | 12 weeks
  The types of repigmentation patterns were classified as perifollicular, marginal, diffuse and mixed configuration.
Transepidermal water loss | 12 weeks
  TEWL at baseline and 12-week's follow-up between 2 groups
Adverse events | 12 weeks
  allergic reactions, edema, erythema, pruritis

CONTACTS AND LOCATIONS:
Overall Officials: Juan Du, Doctor, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking university people's hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No